CLINICAL TRIAL: NCT03693807
Title: A Pilot Protocol Evaluating Safety of Using the Medtronic Pump and Codman Catheter for the Delivery of Hepatic Arterial Infusion (HAI) Chemotherapy in Patients With Colorectal Carcinoma or Cholangiocarcinoma
Brief Title: A Study of the Use of the Medtronic Pump and Codman Catheter to Give Chemotherapy to Patients With Colorectal Carcinoma or Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-343
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; Cholangiocarcinoma
Keywords: Medtronic Pump; Codman Catheter; Hepatic Arterial Infusion (HAI); Floxuridine (FUDR); Gemcitabine; Oxaliplatin; Irinotecan (CPT-11); Fluorouracil; Leucovorin Calcium (Folinic Acid); Dexamethasone; 18-343
MeSH Terms: conditions — Colorectal Neoplasms; Cholangiocarcinoma | interventions — Floxuridine; Gemcitabine; Oxaliplatin; Irinotecan; Fluorouracil; Panitumumab; Cetuximab

STUDY DESIGN:
Intervention Model Description: Pilot non- randomized safety study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Pump Therapy (Experimental): All patients will undergo surgery to have the Medtronic pump and Codman catheter placed appropriately before HAI therapy can begin.
  Interventions: Device: Medtronic pump and Codman catheter; Drug: Floxuridine (FUDR); Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Irinotecan (CPT-11); Drug: Fluorouracil; Drug: Anti-EGFR (Panitumumab or Cetuximab)

INTERVENTIONS:
Device: Medtronic pump and Codman catheter — All patients will undergo surgery to have the Medtronic pump and Codman catheter placed appropriately before HAI therapy can begin.
Drug: Floxuridine (FUDR) — Please see Detailed Description.
Drug: Gemcitabine — Please see Detailed Description.
Drug: Oxaliplatin — Please see Detailed Description.
Drug: Irinotecan (CPT-11) — Please see Detailed Description.
Drug: Fluorouracil — Please see Detailed Description.
Drug: Anti-EGFR (Panitumumab or Cetuximab) — Please see Detailed Description.

SUMMARY:
This study is being done to answer the following question:

Is the combination of the Medtronic pump and the Codman catheter device a safe alternative to the C3000 Codman pump for delivering chemotherapy directly into the liver of patients with metastatic colorectal cancer or cholangiocarcinoma?

DETAILED DESCRIPTION:
Group 1 unresectable liver metastases from colorectal cancer

- Patients will receive either FOLFIRI, FOLFOX, Irinotecan or Irinotecan/oxaliplatin (anti- EGFR agent may be added to any of the systemic treatments) on Days 1 and 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement, so the first doses of systemic chemotherapy will be given on Cycle 1, Day 15, and then every 2 weeks thereafter. CT C/A/P every 2 months. A window of +/- 3 weeks for scans is allowed in order to accommodate patient schedules.

Group 2 resectable liver metastases from colorectal cancer

- Patients will receive either FOLFIRI, FOLFOX, Irinotecan or Irinotecan/oxaliplatin on Days 1 and 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement, so the first doses of systemic chemotherapy will be given on Cycle 1, Day 15, and then every 2 weeks thereafter. Treatment will continue for 6 months in the absence of toxicity or patient withdrawal. CT C/A/P every 3 months. A window of +/- 3 weeks for scans is allowed in order to accommodate patient schedules.

Group 3 unresectable cholangiocarcinoma

- Patients will receive Gemcitabine (800 mg/m2 IV over 30 minutes) and Oxaliplatin (85 mg/ m2 IV over 120 minutes) or Gemcitabine (1000 mg/m2 IV over 30 minutes) alone on Days 1 and 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement, so the first doses of systemic chemotherapy will be given on Cycle 1, Day 15, and then every 2 weeks thereafter. A CT C/A/P every 2 months during treatment. A window of +/- 3 weeks for scans is allowed in order to accommodate patient schedules.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed colorectal adenocarcinoma metastatic to the liver with no clinicalyl or radiographically confirmed extrahepatic disease (or) Histologically confirmed cholangiocarcinoma (Clinical or radiographic evidence of metastatic disease that has been resected is allowed, provided there is no recurrence in that area prior to protocol consent)
* Confirmation of diagnosis must be performed at MSKCC
* Patient may have completely resected hepatic metastases without current evidence of other metastatic disease
* Lab values ≤14 days prior to registration:

  * WBC ≥2.5 K/uL
  * Platelets ≥100,000/uL
  * Creatinine <1.7mg/dL
  * HGB ≥ 8.5 gm/dL
  * Total Bilirubin ≤1.5 mg/dl
* Prior chemotherapy is acceptable if last dose given ≥3 weeks prior to registration to this study. [Note: no chemotherapy to be given after resection of liver lesions prior to treatment on this study]
* Any investigation agent is acceptable if administered ≥3 months before planned first dose on this protocol
* KPS ≥60%
* Patients ≥18 years of age

Exclusion Criteria:

* Prior radiation to the liver (prior radiation therapy to the pelvis is acceptable if competed at least 4 weeks prior to the planned first dose of treatment on protocol)
* Active infection, ascites, hepatic encephalopathy
* Female patients who are pregnant or lactating - or planning to become pregnant within 6 months after the end of the treatment (female patients of child-bearing potential must have negative pregnancy test ≤72 hours before treatment start)
* If in the opinion of the treating investigator a patient has any serious medical problems which may preclude receiving this type of treatment
* Patients with current evidence of hepatitis A, B, C (i.e., active hepatitis)
* Patients with history or known presence of primary CNS tumors, seizures not well-controlled with standard medical therapy, or history of stroke will also be excluded
* Serious or non-healing active wound, ulcer, or bone fracture
* History of other malignancy, except:

  1. Malignancy treated with curative intent and with no known active disease present for ≥3 years prior to registration and felt to be at low risk for recurrence by the treating physician
  2. Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated cervical carcinoma in situ without evidence of disease

There is no exclusion of patients based on sex, ethnicity or race. For these reasons, the study results are expected to be generalizable to the Medicare beneficiary population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kemeny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Unresectable Liver Metastases From Colorectal Cancer; Group 2: Resectable Liver Metastases From Colorectal Cancer; Group 3: Unresectable Cholangiocarcinoma: All patients will undergo surgery to have the Medtronic pump and Codman catheter placed appropriately before HAI therapy can begin.
  Floxuridine (FUDR): Please see Detailed Description.
  Gemcitabine: Please see Detailed Description.
  Oxaliplatin: Please see Detailed Description.
  Irinotecan (CPT-11): Please see Detailed Description.
  Fluorouracil: Please see Detailed Description.
  Anti-EGFR (Panitumumab or Cetuximab): Please see Detailed Description.
Period: Overall Study
Arm/Group | Group 1: Unresectable Liver Metastases From Colorectal Cancer | Group 2: Resectable Liver Metastases From Colorectal Cancer | Group 3: Unresectable Cholangiocarcinoma
Started | 15 | 16 | 4
Completed | 11 | 13 | 2
Not Completed | 4 | 3 | 2
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Unresectable Liver Metastases From Colorectal Cancer | Group 2: Resectable Liver Metastases From Colorectal Cancer | Group 3: Unresectable Cholangiocarcinoma | Total
Number analyzed (Participants) | 15 | 16 | 4 | 35
Age, Continuous [Mean (Full Range); unit: years] | 53 [32 to 78] | 51 [32 to 69] | 62 [39 to 75] | 53 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 3 | 15
  Male | 8 | 11 | 1 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 5
  Not Hispanic or Latino | 12 | 12 | 3 | 27
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 12 | 12 | 4 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 4 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Requiring Stent Replacements
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Unresectable Liver Metastases From Colorectal Cancer | Group 2: Resectable Liver Metastases From Colorectal Cancer | Group 3: Unresectable Cholangiocarcinoma
Number analyzed (Participants) | 15 | 16 | 4
Participants
  Participants requiring stent replacement | 1 | 2 | 1
  Participants not requiring stent replacement | 14 | 14 | 3

2. Primary Outcome: Number of Participants With Any Grade Liver Toxicity
Description: Alkaline phosphatase, serum bilirubin of any patient that received 2 cycles of pump therapy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Unresectable Liver Metastases From Colorectal Cancer | Group 2: Resectable Liver Metastases From Colorectal Cancer | Group 3: Unresectable Cholangiocarcinoma
Number analyzed (Participants) | 15 | 16 | 4
Participants
  Participants with any grade liver toxicity | 12 | 13 | 3
  Participants without any grade liver toxicity | 3 | 3 | 1

3. Secondary Outcome: Overall Survival at 1 Year Assessed as the Number of Participants Who Were Alive or Dead at 1 Year
Description: Overall survival is defined as the time from treatment initiation till the day of death or last follow-up whichever occurs first.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Unresectable Liver Metastases From Colorectal Cancer | Group 2: Resectable Liver Metastases From Colorectal Cancer | Group 3: Unresectable Cholangiocarcinoma
Number analyzed (Participants) | 15 | 16 | 4
Participants
  Alive | 2 | 9 | 1
  Dead | 13 | 7 | 3

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from treatment initiation till the day of progression or death whichever occurs first. Patients that are alive without progression at the end of the study will be censored.
Time Frame: up to 3 years
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Unresectable Liver Metastases From Colorectal Cancer | Group 2: Resectable Liver Metastases From Colorectal Cancer | Group 3: Unresectable Cholangiocarcinoma
Number analyzed (Participants) | 15 | 16 | 4
days | 231 [49 to 812] | 261 [49 to 812] | 531 [49 to 812]

ADVERSE EVENTS:
Time Frame: 1 year
Description: PI has retired and there has been a delay in disaggregating the data. Results will be updated once the disaggregation is complete.
Arm/Group | Group 1: Unresectable Liver Metastases From Colorectal Cancer | Group 2: Resectable Liver Metastases From Colorectal Cancer | Group 3: Unresectable Cholangiocarcinoma
All-Cause Mortality (participants affected / at risk) | 13/15 | 7/16 | 3/4
Serious Adverse Events (participants affected / at risk) | 13/15 | 7/16 | 3/4
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Unresectable Liver Metastases From Colorectal Cancer (N=15) | Group 2: Resectable Liver Metastases From Colorectal Cancer (N=16) | Group 3: Unresectable Cholangiocarcinoma (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Biliary Obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cardiac disorders - Other, specify - Aneurysm of the hepatic artery (Cardiac disorders) | 1 | 0 | 0
Chest pain - Cardiac (Cardiac disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Edema trunk (General disorders) | 1 | 0 | 0
Fever (General disorders) | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 2 | 1
Infections and infestations - Other, specify - Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0 | 0
Surgical and medical procedures - Other, specify - Catheter Dislodge (Surgical and medical procedures) | 0 | 1 | 0
Surgical and medical procedures - Other, specify - Severed catheter (Surgical and medical procedures) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Death NOS (General disorders) | 13 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT03693807/Prot_SAP_000.pdf